CLINICAL TRIAL: NCT06311760
Title: A Phase I, Randomized, Single-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability, And Pharmacokinetics of AZD0292 Following Single Ascending Dose Administration to Healthy Participants
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of a Single Ascending Dose of AZD0292 In Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: D7700C00001
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Healthy Participants Study
Keywords: Monoclonal antibody

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AZD0292 Dose 1 (Experimental): Participants will receive single dose of AZD0292 dose 1 as IV infusion on Day 1.
  Interventions: Drug: AZD0292
- AZD0292 Dose 2 (Experimental): Participants will receive single dose of AZD0292 dose 2 as IV infusion on Day 1.
  Interventions: Drug: AZD0292
- AZD0292 Dose 3 (Experimental): Participants will receive single dose of AZD0292 dose 3 as IV infusion on Day 1.
  Interventions: Drug: AZD0292
- Placebo (Placebo Comparator): Participants will receive matching placebo to AZD0292 as IV infusion on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD0292 — AZD0292 will be administered as single dose via IV infusion.
  Arms: AZD0292 Dose 1; AZD0292 Dose 2; AZD0292 Dose 3
Drug: Placebo — Placebo will be administered as IV infusion.
  Arms: Placebo

SUMMARY:
This study will assess the safety, tolerability and pharmacokinetics (PK) of AZD0292 following intravenous (IV) administration of single ascending doses to healthy adult participants.

DETAILED DESCRIPTION:
This is a First-time-in-human (FTiH) trial.

Eligible participants will be randomized to receive AZD0292 or Placebo. Participants will receive pre-medication with an antihistamine prior to dosing with the study intervention.

The study will comprise:

1. A Screening Period of maximum 28 days.
2. A Treatment Period
3. A Follow-up Period from Day 3 to Day 16
4. An extended Follow-up Period from Day 17 to Day 61

Participants will be involved in this study for a maximum duration of 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All females must have a negative pregnancy test at screening and on admission to the Clinical Unit.
* Females of childbearing potential must not be lactating and if heterosexually active, must agree to use an approved method of highly effective contraception.
* Have a body mass index (BMI) between 18 and 32 kilograms per meter square (kg/m^2) inclusive and weigh at least 50 kilograms (kg) at screening.

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the principal investigator (PI), may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
* History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the previous 6 months prior to screening as well as individuals with a smoking history of tobacco greater than 5 pack years.
* History of alcohol or drug abuse within the past 2 years that, according to the PI, might affect assessments of safety or ability of participant to comply with all study requirements.
* Any drug therapy within 7 days prior to Day 1 (except contraceptives, HRT, or a single use of acetaminophen, aspirin, antihistamine, or combination OTC product that contains acetaminophen with an antihistamine, or OTC nonsteroidal anti-inflammatory agent at a dose equal to or lower than that recommended on the package). Vitamins and other nutritional supplements that are not newly introduced, that is, have been taken for at least 30 days prior to enrollment, are not exclusionary.
* Positive screen for drugs of abuse, alcohol, or cotinine at screening or on admission to the Clinical Unit.
* Any abnormalities in clinical chemistry, hematology, coagulation, or urinalysis results.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity.
* Receipt of another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days or 5 half-lives (whichever is longer) of the study intervention administration in this study. The period of exclusion begins one month after the final dose.
* Receipt of any vaccine within 7 days prior to study intervention administration or planned receipt within 28 days after study intervention administration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Up to 13 weeks
  The safety and tolerability of AZD0292 following IV administration of single ascending doses to healthy adult participants will be assessed.
Number of Participants with Adverse Events of Special Interest (AESI) | Up to 13 weeks
  The safety and tolerability of AZD0292 following IV administration of single ascending doses to healthy adult participants will be assessed.

SECONDARY OUTCOMES:
Maximum Observed Drug Concentration (Cmax) | From Dosing (Day 1) to end of the study (up to 13 weeks)
  The PK (Cmax) of AZD0292 following IV administration of single ascending doses of AZD0292 to healthy adult participants will be assessed.
Area Under Concentration-Curve from Time Zero to the Last Quantifiable Concentration (AUClast) | From Dosing (Day 1) to end of the study (up to 13 weeks)
  The PK (AUClast) of AZD0292 following IV administration of single ascending doses of AZD0292 to healthy adult participants will be assessed.
Area Under Concentration-Time Curve from Time Zero to Infinity (AUCinfinity) | From Dosing (Day 1) to end of the study (up to 13 weeks)
  The PK (AUCinfinity) of AZD0292 following IV administration of single ascending doses of AZD0292 to healthy adult participants will be assessed.
Number of Participants with Positive Anti-drug Antibodies (ADAs) | From Dosing (Day 1) to end of the study (up to 13 weeks)
  The ADA responses following IV administration of single ascending doses of AZD0292 to healthy adult participants will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via there quest portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure."Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment athttps://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/